CLINICAL TRIAL: NCT02978222
Title: A Randomized Multicenter Phase II Trial to Evaluate the Safety, Efficacy and Immunogenicity of Vaccination With Folate Receptor Alpha Peptides With GM-CSF Versus GM-CSF Alone in Patients With Platinum Sensitive Ovarian Cancer and a Response or Stable Disease to Platinum Therapy
Brief Title: Folate Receptor Alpha Peptide Vaccine With GM-CSF Versus GM-CSF Alone in Patients With Platinum Sensitive Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility analysis did not support continuation of the trial
Sponsor: Marker Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRV-004
Record Dates: First submitted 2016-11-22; First posted 2016-11-30 (Estimated); Results first posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2020-02

CONDITIONS: Platinum Sensitive Ovarian Cancer; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Adjuvants, Pharmaceutic; Granulocyte-Macrophage Colony-Stimulating Factor; Single Person; sargramostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FRα peptide plus adjuvant (GM-CSF) (Experimental): FRα peptide vaccine with GM-CSF adjuvant ID administration monthly for 6 months followed by booster administrations every 3 months for up to 1.5 years
  Interventions: Biological: FRα peptide plus Adjuvant (GM-CSF)
- Adjuvant (GM-CSF) Alone (Placebo Comparator): GM-CSF adjuvant alone ID administration monthly for 6 months followed by booster administrations every 3 months for up to 1.5 years
  Interventions: Drug: Adjuvant (GM-CSF) Alone

INTERVENTIONS:
Biological: FRα peptide plus Adjuvant (GM-CSF) — Intradermal injection FRα peptides, 500μg each - plus GM-CSF 125 μg
  Other Names: TPIV200 with GM-CSF adjuvant
  Arms: FRα peptide plus adjuvant (GM-CSF)
Drug: Adjuvant (GM-CSF) Alone — Intradermal injection 125 μg GM-CSF
  Other Names: Leukine®
  Arms: Adjuvant (GM-CSF) Alone

SUMMARY:
This is a double-blind, randomized, parallel groups Phase II trial. Patients with platinum-sensitive advanced ovarian cancer, defined as a lack of progression by RECIST v1.1 criteria following completion of standard-of-care chemotherapy, including a minimum of 4 cycles of a platinum-containing regimen. Patients will be randomized to either the vaccine regimen with GM-CSF adjuvant or GM-CSF adjuvant alone as a control group. Treatment will be administered as a consolidation therapy within one year of the last administration of platinum, targeting the first remission.

DETAILED DESCRIPTION:
This is a multicenter double-blind controlled randomized Phase II study to evaluate the activity of folate receptor alpha (FRα) peptide vaccine as a consolidation treatment following completion of no less than 4 cycles of a platinum containing regimen in patients with platinum-sensitive, non-mucinous ovarian, fallopian tube or primary peritoneal cancer.

The patients will have demonstrated a tumor response or stable disease upon their last regimen (per RECIST v1.1 and/or CA125 GCIG criteria) prior to enrolment in this study.

Following randomization, patients will be administered TPIV200 with GM-CSF adjuvant or GM-CSF control alone. Patients will have booster doses and tumor assessments done every 12 weeks ± 1 week for up to 1.5 years, until objective disease progression or the patient withdraws consent. Tumor responses will be assessed at the study sites by evaluating tumor images/scans according to RECIST v1.1.

ELIGIBILITY:
Criteria for Inclusion:

1. Female patient ≥ 18 years
2. Willing and able to give informed consent
3. Stage III-IV platinum-sensitive (defined as a lack of progression by RECIST v1.1 criteria following completion of standard-of-care chemotherapy, including a minimum of 4 cycles of a platinum-containing regimen) epithelial ovarian, fallopian tube or primary peritoneal carcinoma in first remission.
4. Histologic documentation of diagnosis of carcinoma is required and the following histologic subtypes are eligible: high grade (grade ≥3+) serous or endometrioid carcinoma, carcinosarcoma, or poorly-differentiated adenocarcinoma, or mixed (including above subtypes only). Note that synchronous serous or endometrioid uterine or fallopian cancers are allowed.
5. The patient must have demonstrated an objective response (PR or CR) or stable disease (SD) with the last chemotherapy prior to enrollment and this response must be stable (without progressive disease) before randomization.
6. Patients must receive their first dose of vaccine within 1 year of completion of their final dose of a chemotherapeutic agent of the platinum-containing regimen
7. Adequate normal organ and marrow function within 14 days prior to first vaccine administration:

   * Absolute neutrophil count > 1.5 x 109/L
   * Platelet > 100 x 109/L
   * Hemoglobin > 9.0 g/dL
   * Serum bilirubin < 1.5 times ULN (unless Gilbert's syndrome without concurrent clinically significant liver disease
   * AST/ALT < 2.5 ULN unless liver metastasis in which case it must be < 5 x ULN
   * Serum creatinine CL > 40 mL/min by Cockcroft-Gault formula.
8. Anti-nuclear antibody (ANA) negative or low-positive institutional range, as determined within 28 days from registration. Intermediate values (usually defined by a titer of ≤1:80, or as indicated by institutional range) are acceptable if there are, in the opinion of the Investigator, no early signs of an autoimmune disease.
9. Female subjects must either be of non-reproductive potential (i.e. post-menopause by history: > 60 years old and no menses for > 12 months naturally or secondary to radiation/chemotherapy; OR serum FSH, LH and estradiol levels in the post-menopausal range; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy), or must have a negative serum pregnancy test upon study entry
10. Life expectancy > 24 weeks
11. ECOG performance status of 0 or 1
12. Formalin fixed, paraffin embedded tumor sample from the primary cancer must be sent for central testing.

Criteria for Exclusion

1. Histology consistent with non-serous, non-endometrioid (i.e. mucinous or clear cell), or low-grade or borderline serous ovarian carcinoma
2. Patients with a history of other cancers (other than non-melanoma skin cancers [i.e. basal or squamous cell]) within the past 3 years.
3. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, targeted therapy, biological/cell therapy, tumor embolization, monoclonal antibodies, other investigational agent) < 28 days prior to the first dose of study drug.
4. Current or prior use of immunosuppressive medication within 28 days prior to the fist dose of study drug with the exception of topical, intranasal or inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
5. Active autoimmune disease requiring therapy within the past 2 years. Note: patients with vitiligo, Grave's disease or psoriasis not requiring systemic treatment within the past 2 years are not excluded.
6. History of hypersensitivity to GM-CSF
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
8. Symptomatic thyroid disease, unless negative for thyroid antibodies (TSH receptor, TPO, thyroglobulin).
9. Subjects who are pregnant or are breast feeding.
10. Subjects who or of reproductive potential, and are either:

    * Not abstinent;
    * Not in an exclusive relationship with a partner who is surgically sterile;
    * Not employing an effective method of birth control.
11. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
12. Symptomatic or uncontrolled brain metastasis requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids
13. Subject with uncontrolled seizures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kenney, MD, Study Director — Marker Therapeutics, Inc.
Locations (18):
- United States (18):
  - UAB Gynecology Oncology, Birmingham, Alabama
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Women's Cancer Research Foundation, Newport Beach, California
  - The Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mt. Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialist, West Palm Beach, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Research Partners, Jackson, Mississippi
  - MidAmerica Division, Inc. c/o Research Medical Center, Kansas City, Missouri
  - University Of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Hematology/Oncology Lenox Hill Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - OHSU, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Tennessee Oncology/Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta A, O'Cearbhaill RE, Block MS, Hamilton E, Konner JA, Knutson KL, Potts J, Garrett G, Kenney RT, Wenham RM; TPIV200 Ovarian Cancer Study Investigators (listed at the end). Vaccination with folate receptor-alpha peptides in patients with ovarian cancer following response to platinum-based therapy: A randomized, multicenter clinical trial. Gynecol Oncol. 2024 Oct;189:90-97. doi: 10.1016/j.ygyno.2024.07.675. Epub 2024 Jul 27. PMID 39068739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject screened for trial 20 Jul 2017 and the last subject enrolled was screened 29Nov2018. Seventeen sites (academic and private clinics) in the United States enrolled and treated patients in the trial. The trial was terminated on 18 Oct 2019, after a blinded analysis by the DSMB determined that the futility requirements were not met. While the trial was terminated on 10/18/2019, the last patient could not return for a final visit/safety evaluation until January 15, 2020.
Pre-assignment Details: Enrolled subjects were only excluded from the trial if it was found that inclusion/exclusion criteria were not met for continued participation.
Period: Overall Study
Arm/Group | FRα Peptide Plus Adjuvant (GM-CSF) | Adjuvant (GM-CSF) Alone
Started | 62 | 58
Completed | 1 | 2
Not Completed | 61 | 56
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 0
Not completed — Disease Progression | 32 | 32
Not completed — Early Study Termination | 24 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FRα Peptide Plus Adjuvant (GM-CSF) | Adjuvant (GM-CSF) Alone | Total
Number analyzed (Participants) | 62 | 58 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 34 | 74
  >=65 years | 22 | 24 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 58 | 120
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 58 | 52 | 110
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 55 | 53 | 108
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 62 | 58 | 120
More than 6 months to last date of platinum therapy [Count of Participants; unit: Participants] | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Time to disease progression or recurrence of ovarian cancer defined as disease progression by RECIST 1.1., disease recurrence, death without progression or CA125 progression
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FRα Peptide Plus Adjuvant (GM-CSF) | Adjuvant (GM-CSF) Alone
Number analyzed (Participants) | 61 | 58
Months | 11.1 [8.1 to NA] — The confidence interval upper bound is not able to be estimated because the Kaplan-Meier curve representing the upper confidence limits of the survival function lies above 0.5 | 10.9 [8.0 to 16.8]

2. Secondary Outcome: Overall Survival (OS)
Description: Death with or without ovarian cancer progression
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FRα Peptide Plus Adjuvant (GM-CSF) | Adjuvant (GM-CSF) Alone
Number analyzed (Participants) | 61 | 58
Months | NA [NA to NA] — Point estimates are not able to be estimates because the Kaplan-Meier does not cross 0.5. Confidence interval upper bounds cannot be estimated because the Kaplan-Meier curve representing the upper confidence limits of the survival function lies above 0.5. Additionally, the confidence interval lower bound for the FRα Peptide Plus Adjuvant (GM-CSF) Alone group cannot be estimated because the Kaplan-Meier curve representing the lower confidence limits of the survival function lies above 0.5. | NA [22.8 to NA] — Point estimates are not able to be estimates because the Kaplan-Meier does not cross 0.5. Confidence interval upper bounds cannot be estimated because the Kaplan-Meier curve representing the upper confidence limits of the survival function lies above 0.5. Additionally, the confidence interval lower bound for the FRα Peptide Plus Adjuvant (GM-CSF) Alone group cannot be estimated because the Kaplan-Meier curve representing the lower confidence limits of the survival function lies above 0.5.

3. Secondary Outcome: Best Overall Response Rate
Description: Best overall response defined as sum of Complete Responses and Partial Responses in the subset of patients with measurable tumor lesions at baseline.
  Best overall response is a binary endpoint and defined as a best overall response of either CR or PR among subjects with measurable lesions at baseline, using RECIST v1.1.
  Disease control rate is the percentage of subjects with a response of CR, PR, or SD or non-CR/non-PR vs PD among subjects with measurable lesions at baseline.
Time Frame: 2 years
Population: Subject in MITT with measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | FRα Peptide Plus Adjuvant (GM-CSF) | Adjuvant (GM-CSF) Alone
Number analyzed (Participants) | 6 | 4
Participants | 0 | 3

4. Secondary Outcome: Disease Control Rate
Description: Disease control rate defined as the sum of Complete Responses, Partial Responses and Stable Disease.
  Best overall response is a binary endpoint and defined as a best overall response of either CR or PR among subjects with measurable lesions at baseline, using RECIST v1.1.
  Disease control rate is the percentage of subjects with a response of CR, PR, or SD or non-CR/non-PR vs PD among subjects with measurable lesions at baseline.
Time Frame: 2 years
Population: Subjects in MITT with measurable lesions at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | FRα Peptide Plus Adjuvant (GM-CSF) | Adjuvant (GM-CSF) Alone
Number analyzed (Participants) | 6 | 4
Participants | 6 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected for two years after the first vaccine administration.
Arm/Group | FRα Peptide Plus Adjuvant (GM-CSF) | Adjuvant (GM-CSF) Alone
All-Cause Mortality (participants affected / at risk) | 1/62 | 1/58
Serious Adverse Events (participants affected / at risk) | 8/62 | 8/58
Other Adverse Events (participants affected / at risk) | 61/62 | 56/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FRα Peptide Plus Adjuvant (GM-CSF) (N=62) | Adjuvant (GM-CSF) Alone (N=58)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Closed Right Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Unspecified (incl) cysts and polyps; ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia-unknown etiology (Infections and infestations) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
oral mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FRα Peptide Plus Adjuvant (GM-CSF) (N=62) | Adjuvant (GM-CSF) Alone (N=58)
abdominal distension (Gastrointestinal disorders) | 5 | 7
abdominal pain (Gastrointestinal disorders) | 12 | 14
consipation (Gastrointestinal disorders) | 4 | 6
diarrhea (Gastrointestinal disorders) | 11 | 5
Nausea (Gastrointestinal disorders) | 9 | 7
vomiting (Gastrointestinal disorders) | 7 | 5
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 3
Fatigue (General disorders) | 13 | 12
injection site reaction (General disorders) | 40 | 22
pyrexia (General disorders) | 4 | 3
sinusitis (Infections and infestations) | 3 | 3
upper respiratory tract infection (Infections and infestations) | 3 | 5
urinary tract infection (Infections and infestations) | 7 | 4
fall (Injury, poisoning and procedural complications) | 2 | 3
white blood cell count decreased (Investigations) | 1 | 3
arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 10
back pain (Musculoskeletal and connective tissue disorders) | 7 | 6
myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
headache (Nervous system disorders) | 5 | 5
insomnia (Psychiatric disorders) | 3 | 4
cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6
alopecia (Skin and subcutaneous tissue disorders) | 3 | 3
pruritus (Skin and subcutaneous tissue disorders) | 6 | 4
rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 8
hypertension (Vascular disorders) | 1 | 4

LIMITATIONS AND CAVEATS:
The trial was stopped due futility. Therefore, results are not for the complete study as designed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT02978222/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT02978222/SAP_001.pdf